CLINICAL TRIAL: NCT00968110
Title: Xolair (Omalizumab) Enhances Oral Tolerance Induction in Milk Allergic Children
Brief Title: Xolair Treatment for Milk Allergic Children
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Stanford University (Other)
Responsible Party: Principal Investigator, John Lee, Instructor in Pediatrics, Harvard Medical School, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Milk-01
Record Dates: First submitted 2009-08-27; First posted 2009-08-28 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-09

CONDITIONS: Milk Allergy
Keywords: Milk Allergy
MeSH Terms: conditions — Milk Hypersensitivity | interventions — Omalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Xolair (Experimental): All patients will receive Xolair treatment for 16 weeks.
  Interventions: Drug: omalizumab

INTERVENTIONS:
Drug: omalizumab — Dosing table established for omalizumab
  Other Names: Xolair

SUMMARY:
This is a pilot feasibility study, using Xolair pretreatment for oral milk desensitization. The major assessment will be safety, and the investigators will evaluate for any type of reaction, including allergic reactions that occur during the course of the study.

DETAILED DESCRIPTION:
Our hypothesis is that pretreatment with anti-IgE mAb will greatly reduce the side effects and allergic reactions that occur during oral desensitization to foods and will enhance the development of oral tolerance in patients with severe milk allergy. Once desensitized to milk, children will be able to tolerate milk in a Double Blind Placebo Controlled Food Challenge.

The study will also evaluate whether Xolair provides a robust durability of tolerance once administration of Xolair is terminated. We will examine the specific immunological mechanisms that mediate oral tolerance in children undergoing oral milk desensitization

The trial will be conducted in three parts: (1) pre-treatment with Xolair for 8 weeks, (2) oral desensitization to cow's milk from weeks 9-16 and continued treatment with Xolair for 8 weeks, and (3) double blind placebo controlled food challenge to milk.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe pediatric cow's milk allergy-sensitive subjects between the ages of 4-18 years old.
* Total IgE >30 kU/L
* Sensitivity to cow's milk allergen will be documented by a positive skin prick test result (see Appendix E for details) and RAST test to cow's milk, with 25 kU/L as a lower limit of eligibility. Patients who do not meet the cow's milk RAST requirement may be eligible for this study if they have a history of a moderate to severe reaction, and if they have recently failed an oral food challenge with milk ordered by their physician.
* All female subjects of child-bearing potential will be required to provide a urine sample for pregnancy testing that must be negative one week before being allowed to participate in the study.
* Subjects must be planning to remain in the study area during the trial.
* Subjects and/or their parents must be trained on the proper use of the Epi-Pen to be allowed to enroll in the study.

Exclusion Criteria:

* No absolute contraindications to allergen skin testing and/or oral ingestion of milk are known. However, the risk of serious systemic anaphylactic reactions to milk suggests a number of preexisting conditions that should be considered relative contraindications. Among those conditions are acute infections, autoimmune disease, severe cardiac disease, and treatment with beta-adrenergic antagonistic drugs (beta-blockers).
* Subjects having a history of severe anaphylaxis to milk requiring intubation or admission to an ICU, frequent allergic or non-allergic urticaria, or history consistent with poorly controlled persistent asthma.
* Total IgE > 2000 IU/mL.
* Subjects with unstable angina, significant arrhythmia, uncontrolled hypertension, chronic sinusitis, or other chronic or immunological diseases that in the mind of the investigator might interfere with the evaluation or administration of the test drug or pose additional risk to the subject e.g. gastrointestinal or gastroesophageal disease, chronic infections, scleroderma, hepatic and gallbladder disease, chronic non-allergic pulmonary disease.
* Subject with an FEV1 or PEF less than 80% predicted (moderate persistent asthma) with or without controller medication (if able to perform the maneuver) at screening, the oral desensitization visit, or food challenge visit.
* Subjects who have received an experimental drug in the last 30 days prior to admission into this study or who plan to use an experimental drug during the study.
* Subjects who are current users of oral, intramuscular, or intravenous corticosteroids, tricyclic antidepressants, or are taking a beta-blocker (oral or topical).
* Subjects routinely using medication that could induce adverse gastrointestinal reactions during the study.
* Subjects refusing to sign the EpiPen Training Form (see Appendix F).
* Pregnant or breast feeding females.
* Subjects with a history of rice and soy allergy.

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
The major goal of this study is to assess the safety of Xolair in young children, and the safety of oral desensitization in patients pretreated with Xolair | week 53

CONTACTS AND LOCATIONS:
Overall Officials: Dale Umetsu, MD, Principal Investigator — Boston Children's Hospital
Locations (2):
- United States (2):
  - Stanford Uneiversity Medical Center, Stanford, California
  - Children's Hosptial Boston, Boston, Massachusetts

REFERENCES:
- [Derived] Bedoret D, Singh AK, Shaw V, Hoyte EG, Hamilton R, DeKruyff RH, Schneider LC, Nadeau KC, Umetsu DT. Changes in antigen-specific T-cell number and function during oral desensitization in cow's milk allergy enabled with omalizumab. Mucosal Immunol. 2012 May;5(3):267-76. doi: 10.1038/mi.2012.5. Epub 2012 Feb 8. PMID 22318492